CLINICAL TRIAL: NCT00829179
Title: Role of RhuMab-E25 in Reducing Exhaled NO in Allergic Asthma
Brief Title: Role of RhuMab-E25 in Reducing Exhaled Nitric Oxide (NO) in Allergic Asthma
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Duke University (Other)
Collaborators: Genentech, Inc. (Industry)
Responsible Party: Principal Investigator, John Sundy, Associate Professor, Duke University
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Basic Science
Other Study IDs: 3403; GCRC 894
Record Dates: First submitted 2009-01-22; First posted 2009-01-26 (Estimated); Results first posted 2009-10-21 (Estimated); Last update posted 2016-02-08 (Estimated); Status verified 2016-01

CONDITIONS: Allergic Asthma
Keywords: Asthma
MeSH Terms: conditions — Asthma | interventions — rhuMAb-E25; Omalizumab

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

INTERVENTIONS:
Drug: RhuMab-E25 — three subcutaneous injections spaced 1 month apart; dose based on subject weight and baseline IgE level.
  Other Names: Omalizumab

SUMMARY:
A single center pilot study to determine the protective effects of RhuMAB-E25 on airway physiology and biology in allergic asthmatics that undergo bronchoprovocation with methacholine.

The primary study objective determines the protective impact of RhuMAB-E25 on airway inflammation as reflected in exhaled nitric oxide (NO) levels in allergic asthmatics.

The secondary objective determines the protective effect of rhuMAB E25 against airway bronchoconstriction as reflected in the Provocative Concentration of methacholine to cause a 20% fall in FEV1(PC20) with methacholine challenge testing.

DETAILED DESCRIPTION:
This is a single center prospective, open-label study. Eligible subjects will undergo two baseline measurements of exhaled Nitric Oxide (NO) before and after methacholine challenge testing at least one week apart. All subjects will receive treatment with RhuMAB-E25 in an open label fashion at day 0, weeks 4 and 8, and undergo methacholine challenge and NO measurement at screening/baseline, weeks 0, 6, and 12. Complete Blood Count (CBC) will be done at screening/baseline, weeks 1, 2, 4, 8, and week 12. For women of childbearing potential, a screening pregnancy test will be done. All statistical analysis will occur at the conclusion of this study.

ELIGIBILITY:
Inclusion Criteria:

* Subjects must be at least 18 years of age,
* Must have an FEV1 of > 70% of predicted,
* Must have evidence of bronchial hyperreactivity to methacholine as defined by a methacholine provocation causing a 20% or greater fall in FEV1 (PC20) < 8 mg/ml
* Use of inhaled steroid is permitted; however, no change in inhaled steroid dosage will be permitted over the duration of study
* Must have a normal platelet count,
* Must be willing to and competent to sign the consent form

Exclusion Criteria:

* Subjects that do not have allergic asthma will be excluded.
* Subjects with ER visits or upper respiratory infections within the last six weeks will be excluded.
* Subjects with tobacco use within the past year or > 10 pack year history of tobacco use will be excluded.
* Subjects with serum IgE levels of less than 30 or greater than 700 Iu/mL will be excluded.
* Subjects that require oral steroid use will be excluded.
* Subjects who weigh < 30 kg or > 150 kg are excluded, and subjects with baseline IgE levels greater than 300 may be excluded, depending on weight
* Pregnant or nursing females will be excluded.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 20 (Actual)
Dates: Start 2002-10; Primary Completion 2004-07 (Actual); Study Completion 2004-07 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: John S Sundy, MD, Principal Investigator — Duke University Medical Director
Locations (1):
- Duke University Medical Center, Durham, North Carolina, United States

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Subjects were recruited from the Pulmonary clinic and the local community from 10/2002 - 07/2004
Pre-assignment Details: The majority of screen failures prior to starting study drug was one of 3 reasons; negative methacholine challenge, IgE, too low, or IgE too high.
Groups:
- RhuMab-E25: Subjects with mild asthma received three doses of study drug subcutaneous injections at one month intervals. Dosing range was 150mg-375mg which was based on baseline IGE and subject body weight.
  Subjects with a baseline Ige above 30 and up to 100 with a body weight between 30 and 150kg would receive a study drug dose of 150 mg. Subjects with an IGE 100-200 and body weight 30 - 150 kg would receive a dose of 225 mg. And up to subjects with an IGE of 600-700 only body weight of 30 - 60 would be included with a dose of 375 mg.
Period: Overall Study
Arm/Group | RhuMab-E25
Started | 20
Completed | 19
Not Completed | 1
Not completed — Withdrawal by Subject | 1

BASELINE CHARACTERISTICS:
Arm/Group | RhuMab-E25
Number analyzed (Participants) | 20
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 20
  >=65 years | 0
Age, Continuous [Mean (Standard Deviation); unit: years] | 31.8 (9.1)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 12
  Male | 8
Region of Enrollment [Number; unit: participants]
  United States | 20

OUTCOME MEASURES:

1. Primary Outcome: Change in Exhaled Nitric Oxide From Baseline to Week 12
Description: The primary outcome measure was the change in exhaled nitric oxide levels between baseline and week 12. 12 week value minus baseline value. (Baseline was -1 week, ie 1 week prior to the start of study drug)
Time Frame: 13 weeks
Measure: Mean (Standard Deviation); unit: parts per billion (ppb)
Arm/Group | RhuMab-E25
Number analyzed (Participants) | 19
parts per billion (ppb) | -11.0 (13.3)
Statistical Analysis 1: Comparison: RhuMab-E25; Test type: Superiority or Other; p = 0.005, Sign test; Difference in Mean = 11.0, Standard Deviation 13.3

ADVERSE EVENTS:
Arm/Group | RhuMab-E25
Serious Adverse Events (participants affected / at risk) | 0/20
Other Adverse Events (participants affected / at risk) | 7/20
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | RhuMab-E25 (N=20)
headache (Nervous system disorders) | 2 (3)
cough (Respiratory, thoracic and mediastinal disorders) | 2 (2)
viral syndrome (Infections and infestations) | 3 (3)

LIMITATIONS AND CAVEATS:
Pilot study with small sample size.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No